CLINICAL TRIAL: NCT05414383
Title: A Prospective Study to Evaluate the Diagnostic Accuracy of Computer-aided Diagnosis (CADx) System in Real-time Characterization of Colorectal Neoplasia
Acronym: CADx
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other); University College, London (Other)
Responsible Party: Principal Investigator, Louis Ho Shing Lau, Assitant Professor, Chinese University of Hong Kong
Other Study IDs: 2022.160
Record Dates: First submitted 2022-06-08; First posted 2022-06-10 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CADx: Histopathology prediction by CADx device
  Interventions: Device: CADx
- Endoscopist: Real-time histopathology prediction by expert and non-expert endoscopists

INTERVENTIONS:
Device: CADx — A novel CADx system for real-time histopathological prediction of colorectal neoplasia, by using non-magnified conventional white-light and image enhanced endoscopy.
  Groups: CADx

SUMMARY:
The investigators hypothesize that a newly developed CADx system will have a higher diagnostic accuracy in predicting histopathology of colorectal neoplasia than both expert and junior endoscopists.

DETAILED DESCRIPTION:
Accurate diagnosis and characterization of colorectal polyps is essential before endoscopic resection. Optical diagnosis by enhanced imaging modality (e.g. Narrow Band Imaging, NBI) allows real-time prediction of histopathology. It can assist endoscopists to select the appropriate technique and differentiate between neoplastic or non-neoplastic polyps. Nevertheless, due to the substantial inter-observer variability, the widespread use was limited.

Recently, artificial intelligence and computer-aided polyp diagnosis (CADx) systems have evolved rapidly. The major limitation was the heterogeneity from different types of imaging modalities. Endocytoscopic images require extra steps for pre-staining and magnification, which are time consuming and operator dependent. As a result, it limits the generalisability and applicability in real-world settings.

A novel CADx system will be developed for real-time histopathological prediction of colorectal neoplasia, by using non-magnified conventional white-light and image enhanced endoscopy (NBI). The diagnostic accuracy of this CADx system will be compared with both expert and junior endoscopists.

ELIGIBILITY:
Inclusion Criteria:

1. They have received colonoscopy for screening, surveillance or symptom investigation;
2. They have endoscopic images and videos captured and stored during colonoscopy which are available to be retrieved;
3. They have histologically proven colorectal neoplasia.
4. Written consent obtained

Exclusion Criteria:

1. Poor quality endoscopic images and videos defined as:

   1. Incomplete visualization of the colorectal neoplasia due to technical reasons (e.g. out-of-focus, motion-blurred or insufficient illumination);
   2. Artifacts due to mucus, air bubbles, stool, or blood.
2. Active gastrointestinal bleeding;
3. Fulminant colitis;
4. Obscured view due to poor bowel preparation;
5. Artificial staining of lesion due to chromoendoscopy.
6. Unable to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with colorectal neoplasia
Sampling Method: Probability Sample
Enrollment: 510 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | During the colonoscopy
  area under receiver operating characteristic curves, AUROC in prediction of final histopathology

SECONDARY OUTCOMES:
Sensitivity | During the colonoscopy
  Sensitivity
Specificity | During the colonoscopy
  Specificity
Positive predictive value | During the colonoscopy
  Positive predictive value
Negative predictive value | During the colonoscopy
  Negative predictive value
Diagnostic time | During the colonoscopy
  Diagnostic time

IPD SHARING:
Plan to Share IPD: No